CLINICAL TRIAL: NCT03918278
Title: A Phase 1b, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-0482 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced/Metastatic Solid Tumors.
Brief Title: A Study of MK-0482 as Monotherapy and in Combination With Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-0482-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0482-001; MK-0482-001 (Other: MSD); 2022-500821-34-00 (Registry Identifier: EU CT); U1111-1278-2766 (Registry Identifier: UTN); 2020-004089-20 (EudraCT Number)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Paclitaxel; Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: MK-0482 Monotherapy (Experimental): Participants receive escalating doses of MK-0482 via intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-0482
- Part 1: MK-0482 + Pembrolizumab Combination Therapy (Experimental): Participants receive escalating doses of MK-0482 via IV infusion + pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-0482; Biological: pembrolizumab
- Part 2: Cohort A (Experimental): Participants with metastatic triple negative breast cancer (TNBC) first line treatment (1L) receive MK-0482 via IV infusion plus pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) up to 35 administrations (up to approximately 2 years) and paclitaxel 90 mg/m^2 via IV infusion until PD or discontinuation.
  Interventions: Biological: MK-0482; Biological: pembrolizumab; Drug: Paclitaxel
- Part 2: Cohort B (Experimental): Participants with recurrent non-operable glioblastoma (GBM) current treatment of second line (2L) receive MK-0482 via IV infusion plus pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-0482; Biological: pembrolizumab
- Part 2: Cohort C (Experimental): Participants with metastatic pancreatic ductal adenocarcinoma (PDAC) (1L) receive MK-0482 via IV infusion plus pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) up to 35 administrations (up to approximately 2 years), Nab-Paclitaxel 125 mg/m^2 via IV infusion and gemcitabine 1000 mg/m^2 via IV infusion until PD or unacceptable toxicity that requires discontinuation.
  Interventions: Biological: MK-0482; Biological: pembrolizumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 2: Cohort D (Experimental): Participants with metastatic soft tissue sarcoma (STS) (2L) receive MK-0482 via IV infusion plus pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle (Q3W) up to 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-0482; Biological: pembrolizumab
- Part 2: Cohort E (Experimental): Participants with metastatic non-squamous non-small cell lung carcinoma (NSCLC) (1L) receive MK-0482 via IV infusion plus pembrolizumab 200 mg via IV infusion plus Pemetrexed 500 mg/m^2 via IV infusion on Day 1 of each 21-day cycle (Q3W) up to 35 administrations (up to approximately 2 years) plus carboplatin with desired dose of area under the curve (AUC) 5 and pemetrexed 500 mg/m^2, both administered via IV infusion, followed by maintenance therapy with pemetrexed 500 mg/m^2 via IV infusion for up to a total of 35 administrations (up to approximately 2 years).
  Interventions: Biological: MK-0482; Biological: pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Biological: MK-0482 — IV infusion
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Part 1: MK-0482 + Pembrolizumab Combination Therapy; Part 2: Cohort A; Part 2: Cohort B; Part 2: Cohort C; Part 2: Cohort D; Part 2: Cohort E
Drug: Paclitaxel — IV infusion
  Other Names: Nov-Onxol; Onxol; Paclitaxel Novaplus; Taxol
  Arms: Part 2: Cohort A
Drug: Nab-paclitaxel — IV infusion
  Other Names: Abraxane
  Arms: Part 2: Cohort C
Drug: Gemcitabine — IV infusion
  Other Names: Gemzar
  Arms: Part 2: Cohort C
Drug: Carboplatin — IV infusion
  Other Names: Paraplatin ®
  Arms: Part 2: Cohort E
Drug: Pemetrexed — IV infusion
  Other Names: Alimta
  Arms: Part 2: Cohort E

SUMMARY:
This is a 2 part study. Part 1 is a dose escalation to determine the safety and tolerability and to establish a preliminary recommended Phase 2 dose (RP2D) dose of MK-0482 administered as monotherapy and in combination with pembrolizumab (MK-3475) in participants with advanced solid tumors for which there is no available therapy which may convey clinical benefit. Part 2 is expansion cohort to determine safety and tolerability of MK-0482 in combination with pembrolizumab with and without chemotherapy in participants with advanced tumor specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 only: Has histologically-or cytologically-confirmed advanced/metastatic solid tumors and have received, been intolerant to, or been ineligible for, all treatments known to confer clinical benefit
* Has measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or Response Assessment in Neuro-Oncology (RANO) for Cohort B as assessed by the local site investigator/radiology
* Has provided an evaluable archival or newly obtained tumor tissue sample
* Part 1, Arm 1 only: Has ≥1 discrete malignant lesions that are amenable to biopsy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 95 days after the last dose of chemotherapy: refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent or agree to use contraception unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and ≥1 of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is using a contraceptive method that is highly effective or is abstinent from heterosexual intercourse as their preferred and usual lifestyle during the intervention period and for at least 180 days after the last dose of chemotherapy or 120 days after the last dose of MK-0482 or pembrolizumab, whichever occurs last
* Part 2 Cohort A, C, and E only: WOCBP must also agree not to donate to others or freeze/store for her own use for the purpose of reproduction during and for at least 180 days after the last dose of chemotherapy
* Has a negative highly sensitive pregnancy test within 72 hours before the first dose of study treatment
* Human immunodeficiency virus (HIV) infected participants must have well controlled HIV on anti-retroviral therapy (ART)
* Has adequate organ function
* Part 2 Cohort A only: 1) Has histologically confirmed locally recurrent inoperable or metastatic triple negative breast cancer (TNBC) 2) Has received no prior systemic therapy for metastatic TNBC 3) Has tumor programmed death ligand 1 (PD-L1) combined positive score (CPS) ≥1
* Part 2 Cohort B only: 1) Has confirmed diagnosis of GBM (isocitrate dehydrogenase (IDH) wildtype per 2021 World Health Organization (WHO) classification of tumors of central nervous system) 2) Has received a standard first-line treatment for GBM including surgery and radiation therapy with or without chemotherapy and evidence of disease recurrence or pression by magnetic resonance imaging (MRI) 3) Has time elapsed from prior treatment as per protocol 4) Has Karnofsky performance status (KPS) ≥ 80 within 7 days before start of study treatment 5) Is neurologically stable 6) Has known status of O6-methylguanine-DNA methyltransferase (MGMT) methylation and isocitrate dehydrogenase (IDH)
* Part 2 Cohort C only: Has histologically confirmed diagnosis of metastatic PDAC and has received no prior systemic therapy for metastatic pancreatic ductal adenocarcinoma (PDAC) including chemotherapy, biological or targeted therapy and has albumin ≥3.0 g/dL
* Part 2 Cohort D only: Has histologically confirmed diagnosis of locally advanced or metastatic soft tissue sarcoma (STS) and has received and progressed after one prior line of systemic treatment for advanced STS. Prior treatment in the (neo)adjuvant setting is not counted as a line of treatment for advanced disease
* Part 2 Cohort E only: Has histologically confirmed diagnosis of Stage IV or recurrent non-operable non-squamous non-small cell lung carcinoma (NSCLC) , has confirmation that epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or c-ros oncogene 1 (ROS1) directed therapy is not indicated as primary therapy and has not received prior systemic treatment for metastatic NSCLC

Exclusion Criteria:

* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years; with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody (mAb) and/or any component of pembrolizumab (MK-3475) or MK-0482
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE)
* Has an active infection requiring systemic therapy
* Has a history of interstitial lung disease
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has known Hepatitis B or C infection
* Has received prior systemic anticancer therapy, definitive radiotherapy, including investigational agents within 4 weeks (2 weeks for palliative radiation) before the first dose of study treatment
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study treatment
* Has received an investigational agent or has used an investigational device 4 weeks prior to start of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has had an allogeneic tissue/solid organ transplant in the last 5 years or has evidence of graft-versus-host disease
* Part 2 only: Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or prior therapy targeting other immune-regulatory receptors or mechanisms
* Part 2 Cohort A only: 1) Has a history of class II-IV congestive heart failure or myocardial infarction within 6 months of start of study treatment 2) Has a known sensitivity to any component of paclitaxel or any of its excipients and 3) Is receiving any medication prohibited in combination with paclitaxel unless medication was stopped within 7 days before the start of study treatment
* Part 2 Cohort B only: 1) Has carcinomatous meningitis 2) Has recurrent tumor 3) Has tumor primarily localized to the brainstem or spinal cord 4) Has presence of multifocal tumor, diffuse leptomeningeal or extracranial disease 5) Has evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan except Grade ≤ Grade I and either post-operative OR stable on at least 2 consecutive MRI scans 6) Requires treatment with moderate or high dose systemic corticosteroids as defined in protocol for at least 3 consecutive days within 2 weeks of start of study treatment and 7) Optune® TTFields within 2 weeks of start of study treatment
* Part 2 Cohort C only: 1) Has a history of class II-IV congestive heart failure, cerebral vascular event, unstable angina, or myocardial infarction within 6 months of the start of study treatment 2) Has symptomatic ascites, and 3) Has a known hypersensitivity to nab-paclitaxel or gemcitabine, or any of their excipients
* Part 2 Cohort E only: 1) Has a diagnosis of small cell lung cancer 2) Has symptomatic ascites or pleural effusion 3)Is currently receiving either strong or moderate inhibitors and/or inducers of CYP3A4 or CYP2C8 that cannot be discontinued for the duration of the study 4) Is unable to interrupt aspirin or other NSAIDs, other than aspirin dose ≤1.3 g/day for a 5-day period 5) Is unable or unwilling to take folic acid or vitamin B12 supplementation, and 6) has a known hypersensitivity to carboplatin or pemetrexed, or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Part 1 only) | Cycle 1 (Up to 21 days)
  DLTs defined as any of the following assessed as treatment (Tx)-related by investigator: Grade (Gr)4 nonhematologic toxicity (T); Gr4 hematologic T lasting ≥7 days, except thrombocytopenia (TCP); Gr4 TCP of any duration; Gr3 TCP associated with clinically-significant bleeding; nonhematologic adverse event (AE) ≥Gr3 in severity, with exceptions; Gr3/4 alanine transaminase (ALT), aspartate transaminase (AST), and/or bilirubin (bili) with exceptions; a protocol-defined elevation of ALT, AST, and bili; Gr3/4 nonhematologic laboratory abnormality if: clinically significant medical intervention is required, leads to hospitalization, persists for >1 week, or results in liver injury with exceptions; Gr3/4 febrile neutropenia; >2 week-delay in starting Cycle 2 due to Tx-related T; Tx-related T resulting in Tx discontinuation during DLT evaluation period; missing >25% of the MK-0482 or any combination component during DLT evaluation period resulting from Tx-related AE; or Gr5 toxicity.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 27 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 24 months
  The number of participants who discontinue study treatment due to an AE will be presented.
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Part 2 only) | Up to approximately 28 days from the start of study intervention
  DLTs defined as any of the following assessed as treatment (Tx)-related by investigator: Grade (Gr)4 nonhematologic toxicity (T); Gr4 hematologic T lasting ≥7 days, except thrombocytopenia (TCP); Gr4 TCP of any duration; Gr3 TCP associated with clinically-significant bleeding; nonhematologic adverse event (AE) ≥Gr3 in severity, with exceptions; Gr3/4 alanine transaminase (ALT), aspartate transaminase (AST), and/or bilirubin (bili) with exceptions; a protocol-defined elevation of ALT, AST, and bili; Gr3/4 nonhematologic laboratory abnormality if: clinically significant medical intervention is required, leads to hospitalization, persists for >1 week, or results in liver injury with exceptions; Gr3/4 febrile neutropenia; >2 week-delay in starting Cycle 2 due to Tx-related T; Tx-related T resulting in Tx discontinuation during DLT evaluation period; missing >25% of the MK-0482 or any combination component during DLT evaluation period resulting from Tx-related AE; or Gr5 toxicity.

SECONDARY OUTCOMES:
Minimum Serum Concentration (Cmin) of MK-0482 When Administered as Monotherapy (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 Cmin (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
Cmin of MK-0482 When Administered in Combination with Pembrolizumab (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 Cmin (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
Maximum Serum Concentration (Cmax) of MK-0482 When Administered as Monotherapy (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 Cmax (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
Cmax of MK-0482 When Administered in Combination with Pembrolizumab (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 Cmax (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
Area Under the Concentration-Time Curve (AUC) of MK-0482 When Administered as Monotherapy (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 AUC (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
AUC of MK-0482 When Administered in Combination with Pembrolizumab (Part 1 only) | At designated time points (Up to approximately 25 months)
  Blood samples will be obtained at designated time points for the assessment of MK-0482 AUC (Cycle 1 Day 1: Predose and at end of administration [within 30 minutes after the end of infusion]; Cycle 1 Days 2, 4, 8 and 15: Once daily; Cycles 2, 4, 6, 8 and every 4 cycles thereafter: Predose and at end of administration [within 30 minutes after the end of infusion]; and at end of treatment/discontinuation [Up to approximately 25 months]). Each cycle is 21 days.
Objective Response Rate (ORR) As Assessed by Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) (Part 2 only) | Up to approximately 25 months
  ORR is defined as the percentage of participants who have a complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 will be presented.
ORR As Assessed by Investigator per Response Assessment in Neuro-Oncology (RANO) (Part 2 only) | Up to approximately 25 months
  ORR is defined as the percentage of participants who have a complete response (CR: Disappearance of all target lesions) or a partial response (PR: sum of products of diameters decreased by ≥50% from baseline value) per RANO criteria. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RANO will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- United States (3):
  - Henry Ford Health System ( Site 0002), Detroit, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0003), Hackensack, New Jersey
  - Next Oncology ( Site 0001), San Antonio, Texas
- Australia (2):
  - Macquarie University ( Site 0033), Macquarie University, New South Wales
  - Alfred Health ( Site 0031), Melbourne, Victoria
- Canada (2):
  - BC Cancer - Vancouver Center ( Site 0010), Vancouver, British Columbia
  - Princess Margaret Cancer Centre ( Site 0011), Toronto, Ontario
- Chile (2):
  - FALP-UIDO ( Site 0100), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0101), Santiago, Region M. de Santiago
- Israel (2):
  - Hadassa Ein Karem Medical Center ( Site 0022), Jerusalem
  - Chaim Sheba Medical Center ( Site 0020), Ramat Gan
- Italy (2):
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica ( Site 0091), Siena, Tuscany
  - Istituto Europeo di Oncologia IRCCS-Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative (, Milan
- South Korea (2):
  - Seoul National University Hospital ( Site 0061), Seoul
  - Asan Medical Center ( Site 0060), Seoul
- Hospital Clinic i Provincial ( Site 0041), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26205&tenant=MT_MSD_9011